CLINICAL TRIAL: NCT02793245
Title: Influence of Patient Characteristics on the Tracheobronchial Anatomy Evaluated by a CT Examination
Brief Title: Patient Characteristics and Tracheobronchial Anatomy
Acronym: Scan-Bronchi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014/25; 2014-A00826-41 (Other: ANSM)
Record Dates: First submitted 2016-05-26; First posted 2016-06-08 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Anatomy
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Studied population (Experimental): Patients will be questioned about their main characteristics (age, gender, height, weight, smoking), they will also perform a simplified a pulmonary function test (if possible).
  Interventions: Other: Questionnaire; Other: Simplified pulmonary function test

INTERVENTIONS:
Other: Questionnaire — Questionnaire on their main characteristics : age, gender, height, weight, smoking
Other: Simplified pulmonary function test

SUMMARY:
The clinical use of double lumen tubes and bronchial blockers requires a thorough knowledge of the tracheobronchial anatomy in order to establish the best choice for the patient. The literature is limited regarding major bronchi dimensions. In addition, the measurement method is not always adequate or properly described and some publications have evaluated only the left bronchial diameter. Computed tomography with 3D reconstruction, technical reference, has been little used.

The project is to conduct a prospective study to compare patient characteristics (age, height, weight, gender, smoking, sign of chronic obstructive pulmonary disease (if available), and dimensions of the trachea and of the main bronchi from CT scans with 3D reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* patients aged at least 18 years
* undergoing a CT scan

Exclusion Criteria:

* hospitalized patients,
* people benefiting from a legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2015-06; Primary Completion 2016-11-21 (Actual); Study Completion 2016-11-21 (Actual)

PRIMARY OUTCOMES:
Relationship between patients' age and the minimum diameter of the left main bronchus | 1 year
  Age (years) and diameter (mm)
Relationship between patients' gender and the minimum diameter of the left main bronchus | 1 year
  Gender (male/female) and diameter (mm)
Relationship between patients' height and the minimum diameter of the left main bronchus | 1 year
  Height (cm) and diameter (mm)
Relationship between patients' weight and the minimum diameter of the left main bronchus | 1 year
  Weight (kg) and diameter (mm)

SECONDARY OUTCOMES:
Relationship between patients functional test and the minimum diameter of the left main bronchus | 1 year
  Forced expiratory volume (% of reference value) and diameter (mm)
Relationship between patient characteristics and the measurement of lengths, diameters and cross-sectional areas of the trachea and of right main bronchus | 1 year
Validation of automatic measurement of tracheal and bronchial diameters | 1 year
  Comparison between manual and automatic measurement using the software "Thoracic VCAR" of General Electric

CONTACTS AND LOCATIONS:
Overall Officials: Virginie Dumans-Nizard, MD, Principal Investigator — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jit H, Jit I. Dimensions & shape of the trachea in the neonates, children & adults in northwest India. Indian J Med Res. 2000 Jul;112:27-33. PMID 11006658
- [Background] Chunder R, Nandi S, Guha R, Satyanarayana N. A morphometric study of human trachea and principal bronchi in different age groups in both sexes and its clinical implications. Nepal Med Coll J. 2010 Dec;12(4):207-14. PMID 21744760
- [Background] Zahedi-Nejad N, Bakhshayesh-Karam M, Kahkoei S, Abbasi-Dezfoully A, Masjedi MR. Normal dimensions of trachea and two main bronchi in the Iranian population. Pol J Radiol. 2011 Oct;76(4):28-31. PMID 22802851
- [Background] Benumof JL, Partridge BL, Salvatierra C, Keating J. Margin of safety in positioning modern double-lumen endotracheal tubes. Anesthesiology. 1987 Nov;67(5):729-38. doi: 10.1097/00000542-198711000-00018. PMID 3674473
- [Background] Robinson CL, Muller NL, Essery C. Clinical significance and measurement of the length of the right main bronchus. Can J Surg. 1989 Jan;32(1):27-8. PMID 2642720
- [Background] Eberle B, Weiler N, Vogel N, Kauczor HU, Heinrichs W. Computed tomography-based tracheobronchial image reconstruction allows selection of the individually appropriate double-lumen tube size. J Cardiothorac Vasc Anesth. 1999 Oct;13(5):532-7. doi: 10.1016/s1053-0770(99)90003-4. PMID 10527220
- [Background] Olivier P, Hayon-Sonsino D, Convard JP, Laloe PA, Fischler M. Measurement of left mainstem bronchus using multiplane CT reconstructions and relationship between patient characteristics or tracheal diameters and left bronchial diameters. Chest. 2006 Jul;130(1):101-7. doi: 10.1378/chest.130.1.101. PMID 16840389
- [Background] Breatnach E, Abbott GC, Fraser RG. Dimensions of the normal human trachea. AJR Am J Roentgenol. 1984 May;142(5):903-6. doi: 10.2214/ajr.142.5.903. PMID 6609569
- [Background] Kamel KS, Lau G, Stringer MD. In vivo and in vitro morphometry of the human trachea. Clin Anat. 2009 Jul;22(5):571-9. doi: 10.1002/ca.20815. PMID 19544298
- [Background] Klein U, Karzai W, Bloos F, Wohlfarth M, Gottschall R, Fritz H, Gugel M, Seifert A. Role of fiberoptic bronchoscopy in conjunction with the use of double-lumen tubes for thoracic anesthesia: a prospective study. Anesthesiology. 1998 Feb;88(2):346-50. doi: 10.1097/00000542-199802000-00012. PMID 9477054
- [Background] Mrudula C, Krishnaiah M. The study of bronchial tree. International Journal of Pharma and Bio Sciences 2011;2:B166-B172
- [Background] Otoch JP, Minamoto H, Perini M, Carneiro FO, de Almeida Artifon EL. Is there a correlation between right bronchus length and diameter with age? J Thorac Dis. 2013 Jun;5(3):306-9. doi: 10.3978/j.issn.2072-1439.2013.03.12. PMID 23825764
- [Background] Kim JH, Park SH, Han SH, Nahm FS, Jung CK, Kim KM. The distance between the carina and the distal margin of the right upper lobe orifice measured by computerised tomography as a guide to right-sided double-lumen endobronchial tube use. Anaesthesia. 2013 Jul;68(7):700-5. doi: 10.1111/anae.12208. Epub 2013 May 8. PMID 23656604